CLINICAL TRIAL: NCT04302974
Title: Cohort Study to Investigate the Outcomes of Patients With Hypertension and/or Diabetes Mellitus and the Effectiveness and Cost-effectiveness of Structured Multi-disciplinary Intervention Programmes
Brief Title: Cohort Study on Patient Outcomes, Effectiveness and Cost-effectiveness of Intervention Programmes for DM/HT Patients
Acronym: TRACC
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Danny D. B. Ho Professor in Family Medicine Head, Department of Family Medicine and Primary Care, The University of Hong Kong
Other Study IDs: UW19-329
Record Dates: First submitted 2020-03-03; First posted 2020-03-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Hypertension; Diabetes Mellitus; Cardiovascular Diseases; Morbidity, Multiple; Kidney Disease, Chronic; Death
Keywords: Continuity of care; Multi-morbidity; Effectiveness; Cost-effectiveness; Multi-disciplinary intervention programme
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Cardiovascular Diseases; Renal Insufficiency, Chronic; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Sub-study 1: Trajectory study: All HA primary care patients aged 18 years or above with doctor-documented HT and/or DM receiving care in HA General Out-patient Clinics or Family Medicine Clinics (FMC) identified from the HA CMS database between 2006 and 2019, to explore the trajectory patterns for clinical, treatment and complication profiles and investigate the impact of multi-morbidity, continuity-of-care, different service delivery models and management strategies (including investigation frequency and specific drug regimens) on outcomes and health service utilization.
  Interventions: Procedure: Different structures and processes of primary care management strategies
- Sub-study 2: RAMP-DM: A cohort of patients with i) diagnosis of DM without any known complications on or before September 2010 and ii) Documented management in the HA General Out-Patient Clinics (GOPC) and Family Medicine Clinics (FMC) identified from the HA CMS database between 2009 and 2019, who attended the first RAMP-DM assessment between August 2009 to September 2010
  Interventions: Procedure: Multi-disciplinary Risk Factor Assessment and Management Programmes for diabetes (RAMP-DM)
- Sub-study 2: usual care only: A cohort of patients with i) diagnosis of DM without any known complications on or before September 2010 and ii) Documented management in the HA General Out-Patient Clinics (GOPC) and Family Medicine Clinics (FMC) identified from the HA CMS database between 2009 and 2019, who have never attended any RAMP-DM assessment between August, 2009 to December, 2019
- Sub-study 3: RAMP-HT: A cohort of patients with i) diagnosis of HT without DM and any known complications on or before March 2013 and ii) Documented management in the HA General Out-Patient Clinics (GOPC) and Family Medicine Clinics (FMC) identified from the HA CMS database between 2011 and 2021, who attended the first RAMP-HT assessment between October 2011 to March 2013
  Interventions: Procedure: Multi-disciplinary Risk Factor Assessment and Management Programmes for hypertension (RAMP-HT)
- Sub-study 3: usual care only: A cohort of patients with i) diagnosis of HT without DM and any known complications on or before March 2013 and ii) Documented management in the HA General Out-Patient Clinics (GOPC) and Family Medicine Clinics (FMC) identified from the HA CMS database between 2011 and 2021, who have never attended any RAMP-HT assessment between October 2011 to December 2021
- Sub-study 4: PSCC: A cohort of patients with i) diagnosis of DM without any known complications on or before August 2016, ii) Documented management in the HA General Out-Patient Clinics (GOPC) and Family Medicine Clinics (FMC) identified from the HA CMS database between 2012 and 2021 iii) attended the first RAMP-DM assessment between September, 2012 to August, 2016, who have received the first PSCC call between September, 2012 to August, 2016 after the first RAMP-DM assessment
  Interventions: Procedure: Patient Support Call Centre (PSCC)
- Sub-study 4: without PSCC: A cohort of patients with i) diagnosis of DM without any known complications on or before August 2016, ii) Documented management in the HA General Out-Patient Clinics (GOPC) and Family Medicine Clinics (FMC) identified from the HA CMS database between 2012 and 2021 iii) attended the first RAMP-DM assessment between September, 2012 to August, 2016, who have never received any PSCC services between September 2012 to December 2021

INTERVENTIONS:
Procedure: Different structures and processes of primary care management strategies — Different structures and processes of primary care management strategies includes: Multi-morbidity, continuity-of-care, different service delivery models and management strategies (i.e. investigation frequency and specific drug regimens)
  Groups: Sub-study 1: Trajectory study
Procedure: Multi-disciplinary Risk Factor Assessment and Management Programmes for diabetes (RAMP-DM) — Under the Multi-disciplinary Risk Factor Assessment and Management Programmes (RAMP) for diabetes (RAMP-DM), multi-disciplinary teams of health care professionals (doctors, nurses, dietitians, pharmacists, opticians etc) were established at designated GOPCs. All DM patients are eligible to enrol into the DM RAMP programmes. Each patient in the RAMP receives a comprehensive risk factor and complication screening to determine his/her overall cardiovascular risk and presence of modifiable risk factors, and according to their risk level and need, the patient may receive additional interventions such as additional counselling by the nurse or additional consultations with a senior doctor.
  Groups: Sub-study 2: RAMP-DM
Procedure: Multi-disciplinary Risk Factor Assessment and Management Programmes for hypertension (RAMP-HT) — Under the Multi-disciplinary Risk Factor Assessment and Management Programmes (RAMP) for hypertension (RAMP-HT), multi-disciplinary teams of health care professionals (doctors, nurses, dietitians, pharmacists, opticians etc) were established at designated GOPCs. All HT patients are eligible to enrol into the HT RAMP programmes. Each patient in the RAMP receives a comprehensive risk factor and complication screening to determine his/her overall cardiovascular risk and presence of modifiable risk factors, and according to their risk level and need, the patient may receive additional interventions such as additional counselling by the nurse or additional consultations with a senior doctor.
  Groups: Sub-study 3: RAMP-HT
Procedure: Patient Support Call Centre (PSCC) — RAMP Patients can also be referred to the Patient Empowerment Programme(PEP) - a structured self-care education programme delivered by non-governmental organisations(NGOs). If the DM control is suboptimal but the patient is unable to attend the PEP, they may be referred to the Patient Support Call Centre(PSCC) service. PSCC provides individualized telephone counselling by trained nurses. PSCC empowers high-risk DM patients to engage in self-care behaviours by providing regular protocol-led telephone support to advise and reinforce healthy behaviours. Targeted self-care behaviours include self-monitoring, medication management, balanced diet, exercise, risk factor reduction, problem solving and healthy coping. Enrolled patients receive weekly to bi-weekly calls in the first 3 months and additional calls as required for a maximum of 9 months. Subsequent follow-up calls are undertaken to assess self-care behaviours related to the selected goals and to develop a care plan with the patient.
  Groups: Sub-study 4: PSCC

SUMMARY:
Objectives: To determine the outcome trajectories of patients with hypertension (HT) and/or diabetes mellitus (DM), and evaluate the long-term effectiveness and cost-effectiveness of the Risk Assessment and Management Programmes (RAMP) and other primary care services such as Patient Support Call Centre (PSCC) on reducing complications and mortality

Design: Population-based cohort study

Setting: Hospital Authority (HA) primary care clinics Participants: All patients aged ≥18 years with DM or HT managed in HA primary care clinics between 2006 and 2021

Main outcome measures: (1) incidence of DM/HT-related complications (cardiovascular disease, end-stage renal disease, retinopathy, neuropathy and all-cause mortality); (2) service utilization (out-patient clinics, Accident and Emergency and overnight hospitalizations); (3) Incremental cost-effectiveness ratio per complications or all-cause death avoided, and per QALY gained by RAMP or PSCC.

Methods: A naturalistic cohort study (maximum 10-year follow-up) and retrospective data extraction from the HA clinical management system (CMS) database will be conducted to identify and correlate outcome trajectories of HT and/or DM patients with personal, service delivery and process of care factors. Outcomes of propensity score matched cohorts who have and have not participated in the programmes will be compared. Multivariable Cox proportional hazards regression and Poisson/negative binomial regression will be conducted to evaluate the effect of RAMP, PSCC and other primary care services on the risk of complications, mortality and service utilization. Empirical costs and effectiveness data will be used to calculate cost-effectiveness from the provider's perspective.

Significance: Findings will inform how to optimize service delivery for HT/DM patients in Hong Kong

DETAILED DESCRIPTION:
A naturalistic cohort study with a maximum follow-up period of 10 years, and retrospective extraction of relevant data from the HA clinical management system (CMS) database, designed as four sub-studies:-

1. A trajectory study on all HA primary care patients with HT and/or DM receiving care from 2006 to 2019, to explore the trajectory patterns for clinical, treatment and complication profiles and investigate the impact of multi-morbidity, continuity-of-care, different service delivery models and management strategies (including investigation frequency and specific drug regimens) on outcomes and health service utilization.
2. A 10-year effectiveness and cost-effectiveness analysis (CEA) of RAMP-DM. A cohort of RAMP-DM patients will be compared against a propensity score matched cohort of 'usual care' only DM patients to determine the effectiveness and cost-effectiveness of RAMP-DM on reducing complications and mortality and gain in quality adjusted life years (QALY). The optimal criteria and frequency of repeating RAMP-DM will be determined.
3. A 10-year effectiveness and CEA of RAMP-HT. A cohort of RAMP-HT will be compared against a propensity score matched cohort of 'usual care' only HT patients to determine the effectiveness and cost-effectiveness of RAMP-HT on reducing complications and mortality and gain in QALY. The optimal criteria and frequency of repeating RAMP-HT will be determined
4. An evaluation on the effectiveness and cost-effectiveness of PSCC. A cohort of RAMP-DM plus PSCC (RAMP-DM+PSCC) will be compared against a propensity score matched cohort of RAMP-DM only patients to evaluate the effectiveness and cost effectiveness of PSCC on the reduction of complications and mortality and gain in QALY.

ELIGIBILITY:
Inclusion Criteria:

(Trajectory study)

* All patients aged 18 years or above with a documented doctor-diagnosed DM or HT between 2006 and 2019.
* Documented management in the HA GOPC or FMC identified from the HA CM database between 2006 and 2019.

  (10-year CEA study on RAMP-DM)
* Documented diagnosis of DM without any known complications on or before September 2010
* Documented management in the HA GOPC and FMC identified from the HA CMS database between 2009 and 2019,
* Patients who attended the first RAMP-DM assessment between August 2009 to September 2010 for inclusion in the RAMP-DM cohort
* Patients who have never attended any RAMP-DM assessment between August 2009 to December 2019 for inclusion in the usual care only cohort

  (10-year CEA study on RAMP-HT)
* Documented diagnosis of HT without DM and any known complications on or before March 2013
* Documented management in the HA GOPC and FMC identified from the HA CMS database between 2011 and 2021,
* Patients who attended the first RAMP-HT assessment between October 2011 to March 2013 for inclusion in the RAMP-HT cohort
* Patients who have never attended any RAMP-HT assessment between October 2011 to December 2021 for inclusion in the usual care only cohort

  (5-year CEA study on PSCC)
* Documented diagnosis of DM without any known complications on or before August 2016
* Documented management in the HA GOPC and FMC identified from the HA CMS database between 2012 and 2021,
* Patients who attended the first RAMP-DM assessment between September 2012 to August 2016
* Patients who received the first PSCC call between September 2012 to August 2016 after the first RAMP-DM assessment for inclusion in the PSCC cohort
* Patients who have never received any PSCC services between September 2012 to December 2021 for inclusion in the RAMP only cohort

Exclusion Criteria:

(applicable to all sub-studies)

* Non-Chinese
* Patients with documented DM/HT-related complications diagnosed before the date of enrolment
* Medical specialist outpatient attendance before or within the first year of inclusion to study, to exclude subjects who might have developed complications before study enrolment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * All Chinese patients aged 18 years or above with a documented doctor-diagnosed DM or HT between 2006 and 2021.
  * Documented management in the HA GOPC or FMC identified from the HA CM database between 2006 and 2021.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of DM/HT-related complications (cardiovascular disease, end-stage renal disease, retinopathy, neuropathy and all-cause mortality) | 10 years
  The disease are defined by the diagnosis codes International Classification of Primary Care, Second edition or International Classification of Diseases,Ninth Revision, Clinical Modification.
Service utilization rate (out-patient clinics, Accident and Emergency and hospitalizations) | 10 years
  Based on the electronic health record from Hong Kong Hospital Authority
Incremental cost-effectiveness ratio per DM/HT-related complication or all-cause death avoided, and per QALY gained by RAMP or PSCC | 10 years
  The incremental cost-effectiveness ratio (ICER), that is the ratio of the incremental costs of the RAMP group over the incremental effectiveness, will be calculated for each complication event, or death avoided, and per QALY gain.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L.K. Lam, MD, Principal Investigator — Professor and Head of Department of Family Medicine & Primary Care, HKU
Locations (1):
- Department of Family Medicine & Primary Care, LKS Faculty of Medicine, University of Hong Kong, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Wan EYF, Chin WY, Yu EYT, Chen J, Tse ETY, Wong CKH, Ha TKH, Chao DVK, Tsui WWS, Lam CLK. Retrospective cohort study to investigate the 10-year trajectories of disease patterns in patients with hypertension and/or diabetes mellitus on subsequent cardiovascular outcomes and health service utilisation: a study protocol. BMJ Open. 2021 Feb 5;11(2):e038775. doi: 10.1136/bmjopen-2020-038775. PMID 33550225